CLINICAL TRIAL: NCT07179562
Title: Effectiveness of a Motivational Interviewing Program on the Self-Care Levels of Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Motivational Interviewing Program on the Self-Care in Idiopathic Pulmonary Fibrosis
Acronym: MI-IPF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7820
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to the motivational interviewing intervention group (experimental group) and the standard care group (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "motivational interviewing" program (Experimental): The intervention in the experimental group will consist of a Motivational Interviewing (MI) program conducted in accordance with the Motivational Interviewing Treatment Integrity (MITI) guidelines , lasting 6 months and delivered through video calls and an online platform.
  Interventions: Other: "motivational interviewing"
- Standard of care (No Intervention): Patients followed according to clinical practice.

INTERVENTIONS:
Other: "motivational interviewing" — Randomization for "motivational interviewing"
  Arms: "motivational interviewing" program

SUMMARY:
A specific tool developed to measure self-care in patients with Idiopathic Pulmonary Fibrosis (IPF) is the SC-IPFI, which is an adaptation of an already validated instrument for COPD. It is important to assess how motivational interviewing can influence the self-care behaviors of these patients, better evaluate their level of disease management, prevent the risk of exacerbations, and guide educational interventions.

The primary objective of this study is to evaluate the effectiveness of a motivational interviewing program delivered remotely through video calls and digital platforms in improving the levels of self-care maintenance, self-care monitoring, and self-care management in patients with IPF. The study will also assess the effectiveness of the remotely delivered motivational interviewing program on self-efficacy, anxiety, disease-specific quality of life, therapy adherence, cough, dyspnea, exacerbations, and hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic pulmonary fibrosis according to the 2018 guidelines of the American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association,
* Diagnosed with IPF for at least 1 year,
* Aged 18 years or older,
* Able to express willingness and provide consent to participate in the study,
* In possession of a tablet, smartphone, or computer and internet access via mobile or fixed network.

Exclusion Criteria:

* Diagnosed with dementia,
* Unable to speak, read, or write in Italian,
* Legally blind or deaf,
* In advanced stage of disease (receiving oxygen therapy at 10 to 15 liters per minute).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Il Self Care Index for Pulmonary Idiopatic Fibrosis (SC-IPFI) | 6 months
  The SC-IPFI was derived from a similar tool used for COPD and adapted for idiopathic pulmonary fibrosis. The instrument assesses self-care in fibrotic patients using separate scales for the three dimensions of self-care: self-care maintenance, self-care monitoring, and self-care management. Each scale has a standardized score ranging from 0 to 100, with higher scores indicating better self-care.